CLINICAL TRIAL: NCT01800929
Title: Evaluation of Performance and Usability of N6 in the Paediatric Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cochlear, Asia Pacific (Other)
Collaborators: The HEARing Co-operative Research Centre, Melbourne (Unknown); Melbourne Cochlear Implant Clinic, Melbourne (Unknown); The Shepherd Centre, Sydney (Unknown); Hear and Say Centre (Other); The Hearing House, Auckland (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAP5433
Record Dates: First submitted 2012-08-27; First posted 2013-02-28 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Transplants and Implants; Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- N6 (Experimental): The N6 system comprises an investigational sound processor, remote assistant and fitting software
  Interventions: Device: N6
- N5 (Active Comparator): The current commercially-available cochlear implant system Performance of N5 will be compared to performance with N6 using a within-subject design.
  Interventions: Device: N6

INTERVENTIONS:
Device: N6 — Children with N5 will be upgraded to the N6 for a period of up to 2 months to evaluate.

SUMMARY:
The purpose of this study is to evaluate the performance and usability of the N6 system in children with the N5 system.

DETAILED DESCRIPTION:
This study will evaluate the user benefits of the N6 system in the paediatric population currently equipped with N5. The performance and usability of both systems will be evaluated and compared. The performance of the N6 is expected to be at least equivalent to the N5.

Outcome measures:

* City University of New York (CUNY) Sentence Test in quiet and noise
* Consonant-Nucleus-Consonant (CNC) words in quiet
* in-house designed Usability questionnaires of the N6 system (information to be used internally)
* PEACH, TEACH and SELF questionnaires - developed by Ching & Hill (2007). PEACH - The Parents' Evaluation of Aural/oral performance of Children TEACH - The Teachers' Evaluation of Aural/oral performance of Children for teachers SELF - The Child's Self evaluation of aural/oral performance.

Speech perception tests will be administered at baseline, then again three times, two weeks apart with the N6 processor - i.e. week 0, week 2, week 4 & week 6. Total time: 2 months.

Questionnaires will also be given at the same time points, to get baseline information, as well as N6 information

ELIGIBILITY:
Inclusion Criteria:

* Age 5-14 years, currently using N5
* Minimum speech perception ability in noise of 30% at +10 decibels (dB) signal-to-noise ratio (SNR).
* Minimum of 2 years cochlear implant (CI) experience, including at least 6 months experience with their current processor
* Excellent verbal reporters
* Excellent record of attending clinical appointments.
* Attend a regular school,
* English 1st language.
* Excellent record of compliance with habilitation tasks.

Exclusion Criteria:

* Cognitive impairment, or other significant impairment that would impact on their ability to undertake task requirements
* Inability to attend study appointments.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Group usability performance data for N6 versus N5 | Nov 2012-June 2013
  The investigational sound processor, remote assistant and fitting software will be compared to the existing implant system on measures of speech perception and usability in a take-home study.

SECONDARY OUTCOMES:
speech recognition scores in quiet and noise between the two processors | Nov 2012-June 2013
  The CUNY sentences and CNC word lists will be administered in quiet and noise.
Useability questionnaire on the different sound processing features | Nov 2012-June 2013
  An in house questionnaire has been developed where the parent is asked to rank various features of the device, and its usability on a 5-point Likert Scale
Subjective feedback on performance as well as patient preference between the 2 processors | Nov 2012-June 2013
  The PEACH, TEACH and SELF (Ching & Hill, 2007) will be used to collect this information from the parent, teacher and child. These questionnaires have been used in many previous studies.
  In addition, any verbal feedback provided by recipients will be noted on CRFs.
Evaluate the usability of the two systems in a group of children, their carers and their teachers | Nov 2012-June 2013
  The information from the above questionnaires will be used to collectively compare the usability of the child's current processor and the N6 processor.
Clinical recommendations for fitting paediatric recipients with the new processor | Nov 2012-June 2013

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (3):
  - The Shepherd Centre, Sydney, New South Wales
  - Hear and Say Centre, Brisbane, Queensland
  - Melbourne Cochlear Implant Clinic, Melbourne, Victoria
- The Hearing House, Auckland, New Zealand